CLINICAL TRIAL: NCT04565509
Title: Supporting the Health and Well-being of Children With Intellectual and Developmental Disability During COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 202009060; 3P50HD103525-01S1 (NIH)
Record Dates: First submitted 2020-09-24; First posted 2020-09-25 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Covid19; Intellectual Disability; Developmental Disability; Child Development Disorder
MeSH Terms: conditions — COVID-19; Intellectual Disability; Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: A cluster randomized adaptive trial will be conducted. The first phase will randomize the 6 Special School District schools to either a general message or focus/targeted message. Data analysis will occur and then the schools will be randomized to the best message strategy from phase 1 alone or best message plus and augmented message or implementation strategy.
  The same process will take place independently at the Kennedy Krieger Institutes/Sheppard Pratt Schools.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- General Message (Active Comparator): In phase 1, three schools will be randomized to a messaging strategy that is developed from focus groups that generally describes COVID-19 and the importance of testing.
  Interventions: Behavioral: General Communication Message
- Focus/Targeted Message (Active Comparator): In phase 1, three schools will be randomized to a messaging strategy that is developed from focus groups that is targeted to address specific concerns of the different communities. Messages may target groups being tested (staff versus students) or sociodemographic or race/ethnicity differences between schools depending on the FG input.
  Interventions: Behavioral: Focused/Targeted Message
- Best Message Alone (Active Comparator): In phase 2, the schools will be randomized a second time after data analysis at 5 months to determine which communication strategy is determined to provide the best uptake of testing by students and staff. Three schools will be randomized to receive the best messaging strategy alone to begin at 7 months after testing starts.
  Interventions: Behavioral: Best Message Alone
- Best Message + Augmented Message or Implementation Strategy (Active Comparator): In phase 2, the schools will be randomized a second time after data analysis at 5 months to determine which communication strategy is determined to provide the best uptake of testing by students and staff. Three schools will be randomized to receive the best messaging strategy plus an augmented messaging or implementation strategy. The augmented messaging and implementation strategies will be informed by the barriers and facilitators identified based on the CFIR domains and results of focus groups and surveys in Aim 2.
  Interventions: Behavioral: Best Message + Augmented Message or Implementation Strategy

INTERVENTIONS:
Behavioral: General Communication Message — A messaging strategy will be developed from focus groups that generally describes COVID-19 and the importance of testing.
  Arms: General Message
Behavioral: Focused/Targeted Message — A messaging strategy that is developed from focus groups that is targeted to address specific concerns of the different communities. Messages may target groups being tested (staff versus students) or sociodemographic or race/ethnicity differences between schools depending on the focus groups input.
  Arms: Focus/Targeted Message
Behavioral: Best Message Alone — The best message will be either the general or focused/targeted message described above.
  Arms: Best Message Alone
Behavioral: Best Message + Augmented Message or Implementation Strategy — The augmented messaging and implementation strategies will be informed by the barriers and facilitators identified based on the CFIR domains and results of focus groups and surveys in Aim 2.
  Arms: Best Message + Augmented Message or Implementation Strategy

SUMMARY:
The primary goal of this project is to identify the best messaging and implementation strategies to maximize SARS-CoV-2 testing for children with intellectual and developmental disabilities (IDD) and their teachers to help ensure a safe school environment. Additionally, we will understand nationally the perceptions of COVID-19 and identify facilitators and barriers to help with the adoption of testing in other parts of the US and the necessary strategies to address other mitigation strategies including vaccination.

DETAILED DESCRIPTION:
This research study will occur at six schools dedicated to children with IDD that are a part of the Special School Districts in St. Louis, MO.

Additionally, surveys, focus groups, and fuzzy cognitive mapping sessions will be conducted at these six schools and at schools within the Kennedy Krieger School Programs in Baltimore, MD. Finally, a national survey will be administered to families, teachers, and staff of the 67 University Centers for Excellence in Developmental Disabilities (UCEDD) which is sponsored by the Association of University Centers for Disability (AUCD).

The first aim will involve focus groups of parents/guardians, teachers, and school staff to identify the barriers and facilitators to frequent SARS-CoV-2 testing, impressions of COVID-19, and best messages and implementation strategies to promote increase testing and vaccination. A formal process for developing two types of messages (general versus focused) will be performed using focus group data and involving key stakeholders to test the messages. A cluster randomized adaptive clinical trial will then occur at the six special school district schools. In phase 1, the schools will be randomized initially to either the general or focused message to promote the adoption of weekly SARS-CoV-2 testing by the students and teachers. After 5 months, data analysis will be conducted to determine which strategy led to the highest percentage of testing. Phase 2 will begin at 7 months after the schools are randomized to either the best message determined from phase 1 or best message plus an augmented implementation strategy.

Beginning in April 2021 the first aim was expanded to include weekly testing and message development at the Kennedy Krieger Institutes and Sheppard Pratt Schools in Baltimore, MD. In phase 1, these schools will be randomized initially to either the general or focused message to promote the adoption of weekly SARS-CoV-2 testing by the students and teachers. After 5 months, data analysis will be conducted to determine which strategy led to the highest percentage of testing. Phase 2 will begin at 7 months after these schools are randomized to either the best message determined from phase 1 or best message plus an augmented implementation strategy.

The second aim will assess the national perspectives among parents of children with IDD and school staff regarding the impact of COVID-19 and importance of SARS-CoV-2 testing. Fuzzy cognitive mapping (FCM) and the administration of local and national surveys will be used to accomplish this aim. FCM will involve in-person sessions with parents from the schools in aim 1 and Kennedy Krieger Institute/Sheppard Pratt schools in Baltimore, MD for children with IDD. These sessions will help identify the facilitators and barriers SARS-CoV-2 testing and other mitigation strategies including COVID-19 vaccine. Since no accepted measures have been developed for understanding parent and school staff concerns for children with IDD around COVID-19, local (St. Louis and Baltimore) and national surveys will be conducted. Custom surveys will be deployed across two stakeholder groups: parent/guardians and school staff. We will administer the survey at baseline and during the trial across school settings (St. Louis and Baltimore).

A national survey will also be administered across the UCEDDs. Psychometric analysis will be performed to help identify the questions for a national survey at the end of the study period. In addition to the custom surveys, NIH recommended parent-report surveys from the PhenX Toolkit will be used. The surveys to be used include the Psychological Stress Associated with the COVID-19 Crisis Scale and COVID-19 impact questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in the St. Louis Special School District or the Kennedy Krieger Institutes/Sheppard Pratt Schools in Maryland.
* Teachers/Staff working at the St. Louis Special Schools or the Kennedy Krieger Institutes/Sheppard Pratt Schools in Maryland dedicated to teaching children with IDD.

or

* Parents/ of students, teachers and/or staff employed by the St. Louis Special School District or Kennedy Krieger Institute/Sheppard Pratt schools in Maryland or
* Families, teachers, and staff of the 67 University Centers for Excellence in Developmental Disabilities (UCEDD) which is sponsored by the Association of University Centers for Disability (AUCD).

Exclusion Criteria:

* Members of the research team will not be eligible to participate in the focus groups.

Ages: 5 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Adoption of weekly testing by each participant | 52 weeks
  Ratio of the total number test per the number of weeks of analysis (eg. Phase 1 - 20 weeks)

SECONDARY OUTCOMES:
Acceptability of Messaging/Implementation Strategy | 1 year
  The acceptability of each strategy will be assessed with a validated survey of the families and staff prior to the intervention and at the conclusion of the intervention being utilized.
Feasibility of Messaging/Implementation Strategy | 1 year
  The feasibility of each strategy will be assessed with a validated survey of the families and staff prior to the intervention and at the conclusion of the intervention being utilized.
Appropriateness of Messaging/Implementation Strategy | 1 year
  The appropriate of each strategy will be assessed with a validated survey of the families and staff prior to the intervention and at the conclusion of the intervention being utilized.
Number of missed school days by students or work days by staff | 52 weeks
  The total number of days missed by students and staff at the special schools during the 52 weeks of the study will be obtained.
Students and staff positive SARS-CoV-2 virus | 52 weeks
  The percentage of students and staff positive for SARS-CoV-2 virus will be determined
School-based SARS-CoV-2 transmission events | 52 weeks
  Number of possible SARS-CoV-2 transmission events occurring between students and staff within the school setting.

CONTACTS AND LOCATIONS:
Overall Officials: Jason G. Newland, MD, Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - Hugo W. Moser Research Institute at Kennedy Krieger, Inc., Baltimore, Maryland
  - University of Missouri, Kansas City, Missouri
  - Special School District, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Landes SD, Turk MA, Formica MK, McDonald KE, Stevens JD. COVID-19 outcomes among people with intellectual and developmental disability living in residential group homes in New York State. Disabil Health J. 2020 Oct;13(4):100969. doi: 10.1016/j.dhjo.2020.100969. Epub 2020 Jun 24. PMID 32600948
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Zhou G, Lee MC, Atieli HE, Githure JI, Githeko AK, Kazura JW, Yan G. Adaptive interventions for optimizing malaria control: an implementation study protocol for a block-cluster randomized, sequential multiple assignment trial. Trials. 2020 Jul 20;21(1):665. doi: 10.1186/s13063-020-04573-y. PMID 32690063
- [Background] Ross LF, Loup A, Nelson RM, Botkin JR, Kost R, Smith GR, Gehlert S. Nine key functions for a human subjects protection program for community-engaged research: points to consider. J Empir Res Hum Res Ethics. 2010 Mar;5(1):33-47. doi: 10.1525/jer.2010.5.1.33. PMID 20235862
- [Background] Waltz TJ, Powell BJ, Fernandez ME, Abadie B, Damschroder LJ. Choosing implementation strategies to address contextual barriers: diversity in recommendations and future directions. Implement Sci. 2019 Apr 29;14(1):42. doi: 10.1186/s13012-019-0892-4. PMID 31036028
- [Background] Rader B, Astley CM, Sy KTL, Sewalk K, Hswen Y, Brownstein JS, Kraemer MUG. Geographic access to United States SARS-CoV-2 testing sites highlights healthcare disparities and may bias transmission estimates. J Travel Med. 2020 Nov 9;27(7):taaa076. doi: 10.1093/jtm/taaa076. No abstract available. PMID 32412064
- [Background] Lalli MA, Langmade JS, Chen X, Fronick CC, Sawyer CS, Burcea LC, Wilkinson MN, Fulton RS, Heinz M, Buchser WJ, Head RD, Mitra RD, Milbrandt J. Rapid and Extraction-Free Detection of SARS-CoV-2 from Saliva by Colorimetric Reverse-Transcription Loop-Mediated Isothermal Amplification. Clin Chem. 2021 Jan 30;67(2):415-424. doi: 10.1093/clinchem/hvaa267. PMID 33098427
- [Background] Wylie AL, Fourneir J, Casanovas-Massana A, et al. Saliva is more sensitive for SARS-CoV-2 detection in COVID-19 patients than nasopharyngeal swabs. medRxiv. 2020.
- [Background] Silliman Cohen RI, Bosk EA. Vulnerable Youth and the COVID-19 Pandemic. Pediatrics. 2020 Jul;146(1):e20201306. doi: 10.1542/peds.2020-1306. Epub 2020 Apr 28. No abstract available. PMID 32345686
- [Background] Steiner JF. Using stories to disseminate research: the attributes of representative stories. J Gen Intern Med. 2007 Nov;22(11):1603-7. doi: 10.1007/s11606-007-0335-9. Epub 2007 Sep 1. PMID 17763914
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Jetter AJ, Schweinfort W. Building scenarios with Fuzzy Cognitive Mapping: An exploratory study of solar energy. Futures. 2011;43(1):52-66.
- [Derived] Vestal LE, Schmidt AM, Dougherty NL, Rolf L, Newland JG, Mueller NB; COMPASS-T Study Group. COVID-19 Related Facilitators and Barriers to In-Person Learning for Children With Intellectual and Development Disabilities: A Follow-Up. J Sch Health. 2024 Feb;94(2):105-116. doi: 10.1111/josh.13404. Epub 2023 Oct 18. PMID 37853427
- [Derived] Gemmell M, Walsh T, Sherby M, Imbeah A, Bono K, Baldenweck M, Gurnett C, Newland JG. Clusters of SARS-CoV-2 Infection Across Six Schools for Students with Intellectual and Developmental Disabilities. Infect Dis Ther. 2023 Sep;12(9):2289-2294. doi: 10.1007/s40121-023-00855-5. Epub 2023 Sep 13. PMID 37704799
- [Derived] Vestal LE, Schmidt AM, Dougherty NL, Sherby MR, Newland JG, Mueller NB; COMPASS-T Study Group. COVID-19-Related Facilitators and Barriers to In-Person Learning for Children With Intellectual and Development Disabilities. J Sch Health. 2023 Mar;93(3):176-185. doi: 10.1111/josh.13262. Epub 2022 Nov 20. PMID 36404403
- [Derived] Sherby MR, Walsh TJ, Lai AM, Neidich JA, Balls-Berry JE, Morris SM, Head R, Prener CG, Newland JG, Gurnett CA; COMPASS-T Study Group. SARS-CoV-2 screening testing in schools for children with intellectual and developmental disabilities. J Neurodev Disord. 2021 Sep 1;13(1):31. doi: 10.1186/s11689-021-09376-z. PMID 34465306
- [Derived] Sherby MR, Walsh T, Lai AM, Neidich JA, Balls-Berry JE, Morris SM, Head R, Prener C, Newland JG, Gurnett CA; COMPASS-T Study Group. SARS-CoV-2 Screening Testing in Schools for Children with Intellectual and Developmental Disabilities. Res Sq [Preprint]. 2021 Jul 20:rs.3.rs-700296. doi: 10.21203/rs.3.rs-700296/v1. PMID 34312616
- See also: Brown School Evaluation Center at Washington University in St. Louis — https://evaluationcenter.wustl.edu/
- See also: Health Communication Research Laboratory at Washington University in St. Louis — http://hcrl.wustl.edu/
- See also: Intellectual and Developmental Disabilities Research Center at Washington University in St. Louis — http://iddrc.wustl.edu/
- See also: Kennedy Krieger Institute Intellectual and Developmental Disabilities Research Center — https://www.kennedykrieger.org/research/centers-labs-cores/intellectual-and-developmental-disabilities-research-center-iddrc